CLINICAL TRIAL: NCT03924999
Title: Comparison of Complete Decongestive Therapy (CDT) With Intermittent Pneumatic Compression (IPK) for Treatment of Lipedema
Brief Title: Comparison of Complete Decongestive Therapy With Intermittent Pneumatic Compression for Treatment of Lipedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Tuğba Atan, Assoc. Prof., Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-KAEK-062
Record Dates: First submitted 2019-04-22; First posted 2019-04-23 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Lipedema
Keywords: Lipedema; Combined decongestive treatment; Intermittent pneumatic compression
MeSH Terms: conditions — Lipedema | interventions — carbohydrate-deficient transferrin

STUDY DESIGN:
Who Masked: Investigator
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined decongestive treatment & Combined exercise (Experimental): Combined decongestive treatment consists of manual lymphatic drainage and compression bandaging for 5 days a week, for 6 weeks (totally, 30 sessions).
  All participants received 30 minutes aerobic exercise program including treadmill training consisted of a 5-minute warm-up and cool-down period and 25-minute submaximal aerobic exercise 5 days a week, for 6 weeks. Exercise intensity was calculated from the initial 6MWT. Each session was completed with 15 minutes of strengthening and stretching exercises.
  Interventions: Combination Product: Combined decongestive treatment (CDT) & Combined exercise
- Intermittent pneumatic compression & Combined exercise (Experimental): Intermittent pneumatic compression for 5 days a week, for 6 weeks (totally, 30 sessions).
  All participants received 30 minutes aerobic exercise program including treadmill training consisted of a 5-minute warm-up and cool-down period and 25-minute submaximal aerobic exercise 5 days a week, for 6 weeks. Exercise intensity was calculated from the initial 6MWT. Each session was completed with 15 minutes of strengthening and stretching exercises.
  Interventions: Combination Product: Intermittent pneumatic compression & Combined exercise
- Combined exercise (Active Comparator): All participants received 30 minutes aerobic exercise program including treadmill training consisted of a 5-minute warm-up and cool-down period and 25-minute submaximal aerobic exercise 5 days a week, for 6 weeks. Exercise intensity was calculated from the initial 6MWT. Each session was completed with 15 minutes of strengthening and stretching exercises.
  Interventions: Combination Product: Combined exercise

INTERVENTIONS:
Combination Product: Combined decongestive treatment (CDT) & Combined exercise — Combined decongestive treatment consists of manual lymphatic drainage and compression bandaging for 30 sessions.
  Arms: Combined decongestive treatment & Combined exercise
Combination Product: Intermittent pneumatic compression & Combined exercise — Intermittent pneumatic compression for 5 days a week, for 6 weeks (totally, 30 sessions).
  Arms: Intermittent pneumatic compression & Combined exercise
Combination Product: Combined exercise — 30 minutes aerobic exercise program including treadmill training consisted of a 5-minute warm-up and cool-down period and 25-minute submaximal aerobic exercise 5 days a week, for 6 weeks. Exercise intensity was calculated from the initial 6MWT. Each session was completed with 15 minutes of strengthening and stretching exercises.
  Arms: Combined exercise

SUMMARY:
Lipedema is a chronic, progressive and hereditary adipose tissue disorder characterized by an abnormal increase of subcutaneous adipose tissue, especially in the lower extremities. In contrast to obesity, lipoedema may not improve with weight loss and does not include the risk of metabolic syndrome such as diabetes, hypertension and dyslipidemia. However, if not treated for lipedema, medical complications such as hypermobility, joint problems, walking difficulties, and psychological complications such as anxiety and depression may develop.The aim of this study was to compare the effects of combined decongestive treatment and intermittent pneumatic compression treatment combined with aerobic exercise on pain, quality of life and fatigue in patients with lipedema.

DETAILED DESCRIPTION:
Lipedema is a chronic, progressive and hereditary adipose tissue disorder characterized by an abnormal increase of subcutaneous adipose tissue, especially in the lower extremities. It is often seen in female sex. The main determinants of lipedema are bilateral symmetric swelling of the hypodermis of the legs which are painful with palpation or spontaneous and easy ecchymosis and hematoma with minor trauma.

Lipedema usually begins in the period of hormonal change in adolescence or after a few years and can progress in women during hormone changes such as pregnancy, gynecologic surgery or menopause.

Lipedema is a different diagnosis from obesity, but it can be misdiagnosed as primary obesity due to clinical overlap. In contrast to obesity, lipoedema may not improve with weight loss and does not include the risk of metabolic syndrome such as diabetes, hypertension and dyslipidemia. However, if not treated for lipedema, medical complications such as hypermobility, joint problems, walking difficulties, and psychological complications such as anxiety and depression may develop.

However, if not treated for lipedema, medical complications such as hypermobility, joint problems, walking difficulties and psychological complications such as anxiety and depression may develop.

Treatment for lipedema includes conservative and surgical options. In conservative treatment to control edema, combined decongestive treatment which consists of manual lymphatic drainage and compression bandaging, intermittent pneumatic compression and exercise options are included.

The aim of this study was to compare the effects of combined decongestive treatment and intermittent pneumatic compression treatment combined with aerobic exercise on pain, quality of life and fatigue in patients with lipedema.

ELIGIBILITY:
Inclusion Criteria:

* Subject diagnosed with lipedema according to the criteria of revised Wold.
* Subject did not participate in any exercise program within the last three months.
* No pregnancy / breastfeeding

Exclusion Criteria:

* History of acute infection, cancer, inflammatory rheumatic / connective tissue diseases
* History of cardiovascular or musculoskeletal problems that may prevent them from participating in the exercise program

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female sex
Enrollment: 33 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-12-22 (Actual)

PRIMARY OUTCOMES:
Extremity volumetric measurement | 6 weeks
  Pythagorean theorem in the excel program.
  Pythagorean theorem will automatically calculate volumetric calculation.

SECONDARY OUTCOMES:
Waist circumference | 6 weeks
  Waist circumference
Waist-to-hip ratio | 6 weeks
  Waist-to-hip ratio
6-minute walk test | 6 weeks
  6-Minute Walk Test is a submaximal exercise test usually corresponding to 80% of a subject's maximum heart rate and is used to assess functional capacity and treatment response.
Visual analog scale for pain | 6 weeks
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.
Short Form Health Survey 36 (SF-36) physical performance subscore SF-36 contains 36 items which are used to evaluate the quality of life of patients with chronic pain. | 6 weeks
  Short Form Health Survey 36 (SF-36) physical performance subscore SF-36 contains 36 items which are used to evaluate the quality of life of patients with chronic pain.
Fatigue Severity Scale | 6 weeks
  Fatigue Severity Scale assesses the severity of fatigue during the last week in a 9-item questionnaire (1= strongly disagree, 7= strongly agree). Total score ranges from 9 to 63, with higher scores representing greater fatigue.
Beck Depression Inventory | 6 weeks
  This is a 21-item self-report questionnaire evaluating the presence and severity of depressive symptoms in the vegetative, emotional, cognitive and motivational domains. Scores of each item ranges from 0 to 3, higher scores mean higher risk of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Atan, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reich-Schupke S, Schmeller W, Brauer WJ, Cornely ME, Faerber G, Ludwig M, Lulay G, Miller A, Rapprich S, Richter DF, Schacht V, Schrader K, Stucker M, Ure C. S1 guidelines: Lipedema. J Dtsch Dermatol Ges. 2017 Jul;15(7):758-767. doi: 10.1111/ddg.13036. PMID 28677175
- [Background] WOLD LE, HINES EA Jr, ALLEN EV. Lipedema of the legs; a syndrome characterized by fat legs and edema. Ann Intern Med. 1951 May;34(5):1243-50. doi: 10.7326/0003-4819-34-5-1243. No abstract available. PMID 14830102
- [Background] Canning C, Bartholomew JR. Lipedema. Vasc Med. 2018 Feb;23(1):88-90. doi: 10.1177/1358863X17739698. Epub 2017 Nov 16. No abstract available. PMID 29143577
- [Derived] Atan T, Bahar-Ozdemir Y. The Effects of Complete Decongestive Therapy or Intermittent Pneumatic Compression Therapy or Exercise Only in the Treatment of Severe Lipedema: A Randomized Controlled Trial. Lymphat Res Biol. 2021 Feb;19(1):86-95. doi: 10.1089/lrb.2020.0019. Epub 2020 Dec 9. PMID 33297826